CLINICAL TRIAL: NCT05995067
Title: The Potential Association of Long Non-coding RNA (NEAT1 and MALAT1) in the Process of Epithelial-mesenchymal Transition in Periodontitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ali A Abdulkareem (Other)
Responsible Party: Sponsor-Investigator, Ali A Abdulkareem, assistant professor- department of periodontics-college of dentistry- Baghdad university, University of Baghdad
Organization: University of Baghdad (Other)
Other Study IDs: lncRNA in periodontal disease
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Periodontal Disease, AVDC Stage 3and 4; Epithelial Mesenchymal Transition; Long Noncoding RNA
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — gingival tissue byproduct of resective periodontal surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: -healthy groups/without the condition
- study group: -diseased group-/with the condition (periodontitis)
  Interventions: Other: periodontitis challenge

INTERVENTIONS:
Other: periodontitis challenge — control will be compared to diseased group suffering from periodontal disease.
  Groups: study group

SUMMARY:
Periodontitis is a polymicrobial, inflammatory condition affecting tooth-supporting tissues. It is characterized by a progressive loss of epithelial attachment and resorption of alveolar bone, which can lead to tooth loss. Epithelial-mesenchymal transition (EMT) has been proposed as a reversible process that shifts the cell phenotype from epithelial to mesenchymal-like and may be involved in the process of periodontal inflammation either completely or partially. Long non-coding RNAs (lncRNAs) are a large class of regulatory transcripts longer than 200 nucleotides lacking evident protein-coding potential. Studies have shown that lncRNA dysregulation plays key roles in human diseases, including cancer, by modulating the epithelial-mesenchymal transition (EMT). The involvement of lncRNAs markers in the pathogenesis of periodontal disease induced EMT has not been studied thoroughly and have created a gap in the knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no history of systemic disease e.g., diabetes.
* Both males and females will be included in the study.
* Control group: patients fit the case definition of gingival health2, and confirmed by Histopathological inflammatory cell infiltration analysis.
* Periodontitis group: patients fit the case definition of periodontal disease referred for periodontal flap surgery (modified Widman's flap).
* Patients radiographically confirmed with infrabony pocket eligible for periodontal flap surgery.

Exclusion Criteria:

* Patients not willing to participate or consent.
* Patient taking medications that affect or modify immunity (e.g., corticosteroid), for the last 3 months.
* Patient taking NSAIDs for the last 3 months.
* Active smoker.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with periodontitis, and healthy periodontal tissues will be recruited at the College of Dentistry/University of Baghdad and Al Sadir specialized dental center/Al-Risafa directorate/ Ministry of Health. No age or gender restriction.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
determining the relative expression of lncRNAs (NEAT1 and MALAT1) in healthy and diseased periodontal tissue. | one year
  reverse transcription real time polymerase chain reaction

SECONDARY OUTCOMES:
determine the expression of EMT-related genes (E-cadherin, Vimentin, β-catenin, and Snail1), in healthy and diseased tissues, and their correlation with lncRNAs and clinical parameters. | one year
  reverse transcription real time polymerase chain reaction

CONTACTS AND LOCATIONS:
Locations (1):
- saif mohammed T AL Mufti, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided